CLINICAL TRIAL: NCT00491257
Title: Immunogenicity and Safety of the Inactivated, Split-Virion Influenza Vaccine, Northern Hemisphere 2007-2008 Formulation (Intramuscular Route)
Brief Title: A Study of the Immunogenicity and Safety of the 2007-2008 Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GRT82
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infections
Keywords: Influenza; Orthomyxoviridae Infections; Orthomyxoviruses; Split-virion influenza vaccine
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group 1 (Experimental): Participants aged 18 to 60 years at enrollment
  Interventions: Biological: Inactivated influenza vaccine (split virion) NH 2007-2008 formulation
- Study Group 2 (Experimental): Participants aged 61 years or older at enrollment.
  Interventions: Biological: Inactivated influenza vaccine (split virion) NH 2007-2008 formulation

INTERVENTIONS:
Biological: Inactivated influenza vaccine (split virion) NH 2007-2008 formulation — 0.5 mL, Intramuscular
  Other Names: Vaxigrip

SUMMARY:
This study is designed to generate clinical data as outlined in the Note for Guidance on harmonization requirements for influenza vaccine marketing authorization by the European Medicines Agency.

The objectives of the trial are:

* To determine immunogenicity, of the inactivated, split-virion influenza vaccine Northern Hemisphere (NH) 2007-2008 formulation in terms of the requirements of the Committee for Human Medicinal Products (CHMP) Note for Guidance (NfG) CPMP/BWP/214/96.
* To describe the safety of the inactivated, split-virion influenza vaccine, NH 2007-2008 formulation.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 60 years (i.e. to the day before the 61st birthday) or 61 years or above (from the day of the 61st birthday) on the day of inclusion
* Provision of a signed informed consent
* Able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential: avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination

Exclusion Criteria :

* For a woman of child-bearing potential, known pregnancy or positive urine pregnancy test at Visit 1
* Febrile illness (temperature >= 37.5°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to egg proteins, chicken proteins, or to any of the vaccine components, or history of a life-threatening reaction to the trial vaccine or a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 3 weeks following the trial vaccination
* Previous vaccination against influenza in the previous 6 months
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular vaccination
* Known Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen or Hepatitis C seropositivity
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of 2007-2008 Influenza vaccine (split virion, inactivated). | 21 Days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (2):
- United Kingdom (2):
  - Edinburgh
  - London

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com